CLINICAL TRIAL: NCT03218449
Title: The Prognostic Value of Inflammatory Markers for Postoperative Complications in Patients Undergoing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Brief Title: Inflammatory Markers for Postoperative Complications in Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Yon Hee Shim, Principal Investigator, Gangnam Severance Hospital
Other Study IDs: 3-2017-0053
Record Dates: First submitted 2017-06-22; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/NC: noninfective complication
- 2/IC: infective complication

SUMMARY:
Infective complications after cancer surgery had a significant impact on disease-free and overall survival. Postoperative inflammatory markers have been proven useful in predicting infective complications. However, it remains unknown whether these markers can predict postoperative infection in patients receiving cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) which causes the systemic inflammatory response syndrome. Between September 2014 and April 2017, all patients who underwent cytoreductive surgery and HIPEC for peritoneal carcinomatosis were assessed for postoperative complications. Patients were divided into two groups according to the presence of infective complications. Presence of abscess, positive blood, surgical site, urine or sputum cultures, or clinical signs and symptoms with comparable radiologic findings were defined as infective complications. Retrospectively, C-reactive protein (CRP), neutrophil-to-lymphocyte ratio, white blood cell count, platelet count, mean platelet volume, platelet-to-lymphocyte ratio, albumin were collected from preoperative day and postoperative days (POD) 0-14.

ELIGIBILITY:
Inclusion Criteria:

* Between September 2014 and April 2017, all patients who underwent cytoreductive surgery and HIPEC for peritoneal carcinomatosis

Exclusion Criteria:

* A Patient treated the dexmedetomidine.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between September 2014 and April 2017, all patients who underwent cytoreductive surgery and HIPEC for peritoneal carcinomatosis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
inflammatory markers | up to 2 weeks
  Retrospectively, C-reactive protein (CRP), neutrophil-to-lymphocyte ratio, white blood cell count, platelet count, mean platelet volume, platelet-to-lymphocyte ratio, albumin were collected using electronic medical record from preoperative day and postoperative days (POD) 0-14.

CONTACTS AND LOCATIONS:
Overall Officials: Yon Hee Shim, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea